CLINICAL TRIAL: NCT03934489
Title: Reducing Depression and Anxiety in Individuals With Multiple Sclerosis (MS) and Their Support Partners: An Emotion Regulation Skills Training Intervention
Brief Title: Emotion Regulation Skills Training for Individuals With MS and Their Support Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00199623; PP-1804-30860 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERSIST (Experimental): Participants will receive Partnered Emotion Regulation Skills Intervention and Support.
  Interventions: Behavioral: PERSIST
- Facilitated Peer Support (Active Comparator): Participants will undergo a 12-week group intervention, adapted from community-based peer support groups, that focuses on participant-generated topics and facilitated discussion.
  Interventions: Behavioral: Facilitated Peer Support

INTERVENTIONS:
Behavioral: PERSIST — 12-week group, adapted from Dialectical Behavior Therapy, that focuses on emotion regulation skills training and practice.
  Arms: PERSIST
Behavioral: Facilitated Peer Support — 12-week group, adapted from community-based peer support groups, that focuses on participant-generated topics and facilitated discussion.
  Arms: Facilitated Peer Support

SUMMARY:
This pilot randomized controlled trial investigates a novel, group-based emotion regulation skills training intervention for reducing anxious and depressive symptomatology and improving emotion regulation and problem solving in individuals with MS and the individual's support partners. Participants will be randomized (1:1) to the intervention ("Partnered Emotion Regulation Skills Intervention and Supportive Teaching [PERSIST]") or to the active control (Facilitated Peer Support).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* able to speak/read in English
* able to commit to attending at least 9 of the 12 weekly group sessions
* individuals with MS must be relapse/exacerbation-free for at least 1 month
* support partners must score at least 8 on the HADS-D or HADS-A
* individuals with MS must score a least 11 on the HADS-D or HADS-A

Exclusion Criteria:

* under 18 years old
* unable to speak/read in English
* unable to commit to attending at least 9 of the 12 weekly group sessions
* MS relapse within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Depression Subscale score of the Hospital Anxiety and Depression Scale (HADS-D) | Baseline, 13 and 26 weeks
  The HADS-D is a 7-item subscale of the HADS that measures depressive symptomatology. Scores range from 0 to 21 points (each item is rated 0-4), with higher scores indicating greater depressive symptomatology.
Change in Anxiety Subscale score of the Hospital Anxiety and Depression Scale (HADS-A) | Baseline, 13 and 26 weeks
  The HADS-A is a 7-item subscale of the HADS that measures anxious symptomatology. Scores range from 0 to 21 points (each item is rated 0-4), with higher scores indicating greater anxious symptomatology.

SECONDARY OUTCOMES:
Change in Difficulties in Emotion Regulation Scale (DERS-16) score | Baseline, 13 and 26 weeks
  The DERS-16 is a 16-item self-report measures that assesses difficulties with managing negative emotions, distress, and impulsivity. Scores range from 16 to 80 points (each item is rated 1-5), with higher scores indicating greater emotional dysregulation.
Change in Problem Solving Inventory (PSI) score | Baseline, 13 and 26 weeks
  The PSI is a 32-item self-report instrument designed to assess perceived problem solving abilities. Scores range from 32 to 192 points (each item is rated 1-6), with higher scores indicating greater difficulty with problem solving.
Change in RAND 36-Item Short Form Health Survey (SF-36) score | Baseline, 13 weeks, and 26 weeks
  The SF-36 is a 36-item self-report measure of health-related quality of life. The scale is divided into 8 subscales, each ranging from 0 to 100 points, with higher scores indicating better health-related quality of life.
Change in Zarit Burden Interview (ZBI) score | Baseline, 13 weeks, and 26 weeks
  The ZBI is a 22-item self-report measure of caregiver burden. Scores range from 0 to 88 (each item is rated 0-4), with higher scores indicating greater burden.

CONTACTS AND LOCATIONS:
Overall Officials: Abbey Hughes, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States